CLINICAL TRIAL: NCT01652079
Title: A Phase II, 2-stage Trial of CRLX101 in Combination With Bevacizumab in Recurrent Platinum-Resistant Ovarian, Tubal and Peritoneal Cancer
Brief Title: CRLX101 in Combination With Bevacizumab for Recurrent Ovarian/Tubal/Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Thomas Penson, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-485
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Epithelial; Primary
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — IT-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): CRLX101
  Interventions: Drug: CRLX101

INTERVENTIONS:
Drug: CRLX101 — q 14 days

SUMMARY:
This research study is a Phase II clinical trial. In addition to studying safety, Phase II clinical trials test if the investigational drug is effective and whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved CRLX101 for your type of cancer.

Camptothecin is a chemical extracted from plants that is the basis for the standard FDA-approved chemotherapy drugs irinotecan and topotecan. Camptothecin works by interfering with the way cells divide and multiply. The investigational drug CRLX101 is a formulation of camptothecin and a large molecule (nanoparticle)that appears to allow more of the camptothecin to get into tumors and stay in tumors. The persistence of the CRLX101 in the tumor may increase the probability that the tumor cells will be damaged.

CRLX101 has been well tolerated in the laboratory and in participants with different kinds of cancer.

Bevacizumab (Avastin) is a VEGF inhibitor which has activity in many kinds of cancer. Bevacizumab has been successfully combined with many chemotherapy partners.

It has been hypothesized that the combination of bevacizumab with CRLX101 might have unique clinical activity in combination in the treatment of this disease due to the simultaneous inhibition of distinct steps along the HIF → (CAIX) → VEGF → VEGFR2 pathway. Specifically, it is hypothesized that CRLX101-mediated inhibition of HIF-1α carries with it the potential to interrupt hypoxia and HIF-1α-associated resistance to VEGFR inhibitors. It is hoped that this combination will work to treat your type of cancer.

DETAILED DESCRIPTION:
You will receive CRLX101 and bevacizumab through an intravenous (IV) infusion once every 14 days. Each cycle is 28 days. You will continue to receive both drugs until you and/or the research doctor decides it may not be in your best interest to continue.

You will receive premedication including decadron, zantac and benadryl to help prevent an allergic reaction and nausea prior to your CRLX101 infusion.You will also receive IV fluid before and after the study drug administration to keep you hydrated. It will be important for you to drink water regularly in between study visits.You will be treated as an outpatient. At every clinic visit, you will undergo the following assessments: Medical history, physical examination, vital signs, performance status, routine blood tests, urine tests, assessment for any new side effects, CT evaluation (every 8 weeks).

You will have an end of study visit within 30 days of your last dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian, tubal or primary peritoneal cancer
* Measurable disease
* May have received up to 2 prior cytotoxic chemotherapy
* Life expectancy of greater than 3 months

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior camptothecin, prior VEFG inhibitors
* Gross hematuria
* Chemotherapy or radiotherapy within 4 weeks of study entry
* uncontrolled HTN
* Receiving other study agents
* History of allergic reaction to compounds of similar chemical or biologic composition to topotecan or irinotecan
* Known brain metastases
* History of a different malignancy within the previous 2 years
* Intercurrent illness
* HIV positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months
  Progression free survival at 6 months (PFS6) using RECIST 1.1

SECONDARY OUTCOMES:
Response Rate | 2 years
  Response Rate (CR+PR) using RECIST 1.1
Assessment of Toxicity | 2 years
  Assessment of toxicity
Analysis of biopsies | 2 years
  Analysis of ovarian tumor biopsies and ascites of the presence or absence of CRLX101 or the active drug, camptothecin

CONTACTS AND LOCATIONS:
Overall Officials: Richard Penson, MD, MRCP, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts